CLINICAL TRIAL: NCT06012175
Title: Efficacy and Safety of Melatonin for Pain Relief in Knee Osteoarthritis Patients: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Melatonin for Knee Osteoarthritis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Collaborators: Peking University People's Hospital (Other); West China Hospital (Other); Massachusetts General Hospital (Other); School of Medicine, University of Nottingham (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20230731
Record Dates: First submitted 2023-08-08; First posted 2023-08-25 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Melatonin; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral melatonin supplementation (Experimental): Participants in the intervention arm will receive one 3 mg melatonin tablet every night before going to bed
  Interventions: Dietary Supplement: Melatonin
- Placebo (Placebo Comparator): The control group will receive an identical-looking inert placebo tablet every night before going to bed
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Melatonin — One 3 mg melatonin tablet every night before bedtime for 12 weeks
  Arms: Oral melatonin supplementation
Dietary Supplement: Placebo — One placebo tablet, having an identical appearance to the melatonin tablet, every night before bedtime for 12 weeks
  Arms: Placebo

SUMMARY:
By recruiting knee osteoarthritis patients and treating them with melatonin, this study aims to determine the efficacy and safety of melatonin in alleviating pain in this patient population.

DETAILED DESCRIPTION:
Knee osteoarthritis (KOA) is a major source of pain and disability among adults worldwide, but the treatment options for patients with painful KOA are inadequate. The current first-line oral drugs have only small to moderate benefits, and some may have serious adverse effects. Therefore, it is important to identify novel therapeutic medications with satisfactory efficacy and acceptable side-effect profiles for KOA.

Melatonin (N-acetyl-5-methoxytryptamine), an indolamine mainly secreted in the pineal gland, is generated from the amino acid tryptophan via derivatization reactions. There are numerous experimental and clinical data supporting the analgesic role of melatonin. In experimental studies, melatonin shows potent analgesic effects in a dose-dependent manner. In clinical studies, melatonin has been shown to have analgesic benefits in people with chronic painful conditions, such as fibromyalgia, irritable bowel syndrome, and migraine. In an animal OA study, the investigators found that melatonin reverses pain behaviors and synovial inflammation, and down-regulates pain sensitization-related neuromediators in the synovium. These findings suggest that melatonin may be potentially effective in treating OA-related pain. However, there is a paucity of high-quality clinical evidence from human studies.

The investigators propose to conduct a randomized, double-blind, placebo-controlled trial to examine the efficacy and safety of 12 weeks treatment with oral melatonin on pain and function in patients with KOA.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 40 and 80 years.
2. Knee OA according to the American College of Rheumatology (ACR) clinical criteria.
3. Knee pain lasting 3 months or longer and a score of 7 or greater on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale (standardized to range from 0-20).
4. Kellgren-Lawrence (KL) grade 2 or 3.
5. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Any use of NSAIDs or other analgesics in the past two weeks.
2. History of injections of corticosteroids in the past three months or hyaluronic acid in the past 6 months in the index knee.
3. History of arthroscopy or open surgery in the index knee in the past 12 months.
4. History of a knee replacement in the index knee or planning to receive such a procedure within 3 months.
5. History of a severe injury in the index knee.
6. Pain in the index knee caused by inflammatory, autoimmune, neoplastic diseases or other diseases.
7. Abnormal liver or kidney functions, as defined by alanine transaminase or aspartate aminotransferase >two times the upper limit of normal, or blood urea nitrogen or serum creatinine >two times the upper limit of normal.
8. Severe cardiopulmonary diseases.
9. Uncontrolled hypertension or diabetes mellitus.
10. Diagnosis of malignant tumors.
11. Pregnant or contemplating pregnancy or breastfeeding.
12. Any use of melatonin supplement before enrollment within 30 days.
13. Allergic to melatonin or its preparation.
14. Any use of anti-depressive/psychotropic drugs.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score. | Baseline, Week 12
  WOMAC is a self-administered, disease-specific questionnaire that assesses the severity of OA symptoms. The reliability and validity of WOMAC have been confirmed in many clinical trials. WOMAC subscales consist of pain (5 items), stiffness (2 items), and physical function (17 items). Each item is rated from 0 to 4, totaling scores of 0-20, 0-8, and 0-68 for pain, stiffness, and function subscales, respectively.

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain score. | Baseline, Weeks 2, 4, 6, 8 and 10
  WOMAC is a self-administered, disease-specific questionnaire that assesses the severity of OA symptoms. The reliability and validity of this index have been confirmed in many clinical trials. WOMAC subscales consist of pain (5 items), stiffness (2 items), and physical function (17 items). Each item is rated from 0 to 4, totaling scores of 0-20, 0-8, and 0-68 for pain, stiffness, and function subscales, respectively.
Knee pain on a visual analogue scale (VAS). | Baseline, Weeks 2, 4, 6, 8, 10, and 12
  Knee pain will be assessed by a VAS from 0 to 100, with 0 indicating "No pain" and 100 indicating "Very severe pain".
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) total score. | Baseline, Weeks 2, 4, 6, 8, 10 and 12
  WOMAC is a self-administered, disease-specific questionnaire that assesses the severity of OA symptoms. The reliability and validity of this index have been confirmed in many clinical trials. WOMAC subscales consist of pain (5 items), stiffness (2 items), and physical function (17 items). Each item is rated from 0 to 4, totaling scores of 0-20, 0-8, and 0-68 for pain, stiffness, and function subscales, respectively.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) stiffness score. | Baseline, Weeks 2, 4, 6, 8, 10 and 12
  WOMAC is a self-administered, disease-specific questionnaire that assesses the severity of OA symptoms. The reliability and validity of this index have been confirmed in many clinical trials. WOMAC subscales consist of pain (5 items), stiffness (2 items), and physical function (17 items). Each item is rated from 0 to 4, totaling scores of 0-20, 0-8, and 0-68 for pain, stiffness, and function subscales, respectively.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) function score. | Baseline, Weeks 2, 4, 6, 8, 10 and 12
  WOMAC is a self-administered, disease-specific questionnaire that assesses the severity of OA symptoms. The reliability and validity of this index have been confirmed in many clinical trials. WOMAC subscales consist of pain (5 items), stiffness (2 items), and physical function (17 items). Each item is rated from 0 to 4, totaling scores of 0-20, 0-8, and 0-68 for pain, stiffness, and function subscales, respectively.
Patient global assessment of osteoarthritis (PGA-OA). | Baseline, Weeks 2, 4, 6, 8, 10 and 12
  PGA-OA score will be assessed using a 100 mm visual analogue scale (higher is worse).
SF-12 questionnaire. | Baseline, Weeks 2, 4, 6, 8, 10 and 12
  The SF-12 questionnaire includes 8 multi-item domains (i.e., physical function, social function, role-emotional, role-physical, bodily pain, general health, mental health, and vitality). These can be combined into 2 summary measures (i.e., physical and mental component summary measures).
Hospital Anxiety and Depression Scale (HADS). | Baseline, Weeks 2, 4, 6, 8, 10 and 12
  HADS is a self-report scale comprising 14 items. Of them, 7 evaluate depression and 7 anxiety symptoms. The score of each domain ranges from 0 to 21. The higher scores equal greater involvement of either anxiety or depression.
Pittsburgh Sleep Quality Index (PSQI). | Baseline, Weeks 2, 4, 6, 8, 10 and 12
  PSQI is a self-rated questionnaire that assesses sleep quality and disturbances over a 1-month interval. PSQI consists of 19 self-assessments and is categorized into seven dimensions (quality of sleep, fall asleep, sleeping time, sleep efficiency, sleep disorders, hypnotic medications, and daytime dysfunction). Each dimension scores from 0 to 3 points, and the total score of the PSQI is the sum of points of seven dimensions, ranging from 0 to 21 (higher is worse).
Timed Up and Go Test (TUG). | Baseline, Weeks 4, 8, and 12
  TUG is a functional performance measure specifically for knee and hip OA. TUG directly evaluates an individual's ability to transfer, ambulate and maintain balance during transitions. TUG assesses the time it takes participants to get up from a standard-height chair, walk 3 m, turn and return to the chair, and sit down again. TUG has good interrater and intrarater reliability and validity for functional testing in older adults.
20-m Walk Test. | Baseline, Weeks 4, 8, and 12
  The 20-m walk test has been recommended to assess physical function in individuals with knee OA. Participants will be instructed to walk at their usual walking speed from start to finish points of a marked 20-m distance.
Chair-stand Test. | Baseline, Weeks 4, 8, and 12
  The chair-stand test will use a standard chair with a 47-cm seat height. Participants start the test seated, with arms crossing over the chest, and are instructed to rise to a full stand and return to the initial seated position as many times as possible in 30 s. The total number of completed chair stands is averaged across two trials and used for analysis. A greater number of chair stand repetitions is interpreted as better performance.
Ultrasound-assessed knee synovitis. | Baseline, Week 12
  Both knees will be assessed with the participant supine and the knee in 30° flexion. The suprapatellar bursa will be scanned according to the Outcome Measures in Rheumatology (OMERACT) atlas. Synovial hypertrophy and effusion will be assessed using OMERACT-7 definitions. The maximal synovial thickness and effusion depth will be measured in millimeters using the longitudinal axis. Synovial hypertrophy is defined as synovial thickness ≥4 mm, and joint effusion is defined as depth of effusion ≥4 mm according to the European League Against Rheumatism (EULAR) criteria. Power Doppler signal (PDS) observed in the synovial membrane in both longitudinal and transverse planes will be scored using a semi-quantitative grading system from 0 to 3 (0 = absent, 1 = mild, 2 = moderate, 3 = marked or severe). Participants will be defined as having synovial hypertrophy or PDS if these features are present in either knee.
Rescue medicine consumption. | Weeks 2, 4, 6, 8, 10 and 12
  Patients will be permitted to use acetaminophen as rescue medication, and the consumption of rescue medication will be recorded at each visit and in the daily logs.
C-reactive protein (CRP). | Baseline, Weeks 4, 8, and 12
  The blood samples will be collected in the morning after an overnight fast at baseline and the following visits. to measure the level of CRP in serum.
Microbiota diversity and composition. | Baseline, Weeks 4, 8, and 12
  Stool, and saliva samples will be collected at baseline and the following visits. Microbial diversity will be quantified via the Shannon diversity index, and microbiota composition will be identified on different levels including phylum, family and genus.
Incidence of adverse events and serious adverse events. | Weeks 2, 4, 6, 8, 10 and 12
  Adverse events and serious adverse events will be measured and recorded.

OTHER OUTCOMES:
Short Physical Performance Battery (SPPB) scores. | Baseline, Weeks 4, 8, and 12
  The SPPB is a standardized, reproducible measure of global physical function validated in frail older persons that predicts a wide range of clinical outcomes. It has 3 components: a standing balance test, a gait speed (4-m walk) test, and a strength test (time to complete 5 chair rises). Each component is scored 0-4 for a total score ranging from 0-12, where lower scores indicate more severe physical dysfunction.
Grip strength. | Baseline, Week 4, 8, and 12
  The grip strength of the dominant hand of the participants will be measured using a calibrated Jamar dynamometer with the participants in the sitting position (Patterson Medical, Ltd. Nottinghamshire, UK). Three grip strength measurements will be taken at 10 s intervals, and the maximum value of the three measurements will be used as the participant's final grip strength.
Bone mineral density (BMD). | Baseline, Week 12
  A trained technician will measure the BMD of all participants. The total body BMD and site-specific BMD at the lumbar spine, pelvis, trunk, femoral neck, trochanteric, and ward's triangle, will be all measured. The dual-energy X-ray absorptiometry (DXA) scan results will be reported as absolute values of BMD (g/cm2).
DXA -based whole body muscle mass. | Baseline, Week 12
  The assessment of body composition provides insights into the nutritional status and functional capacity. It helps understanding nutrition in the developmental origins of health and disease and in monitoring therapeutic interventions. The whole body muscle mass will be measured using DXA.
DXA -based whole body fat mass. | Baseline, Week 12
  The assessment of body composition provides insights into the nutritional status and functional capacity. It helps understanding nutrition in the developmental origins of health and disease and in monitoring therapeutic interventions. The whole body fat mass will be measured using DXA.

CONTACTS AND LOCATIONS:
Overall Officials: Chao Zeng, MD, PhD, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No